CLINICAL TRIAL: NCT04162821
Title: Clinical Pharmacokinetics of Hydroxynitone Capsules in Healthy Chinese Subjects
Brief Title: Study on Pharmacokinetics of Hydronidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GNI-F351-201902
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetics of Hydronidone
MeSH Terms: interventions — hydronidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 60mg group (Experimental)
  Interventions: Drug: Hydronidone
- 90mg group (Experimental)
  Interventions: Drug: Hydronidone
- 120mg group (Experimental)
  Interventions: Drug: Hydronidone

INTERVENTIONS:
Drug: Hydronidone — Take hydroxynitone capsule

SUMMARY:
To evaluate the pharmacokinetic characteristics of hydronidone capsules (specification: 30 mg/ pill) in healthy subjects And the effect of feeding on pharmacokinetics to provide evidence for phase II/III clinical trial protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, half male and half female;
2. Age: from 18 to 45 years old, the age difference of the same group of subjects should not be more than 10 years;
3. Weight: male ≥50kg, female ≥45kg, 19≤BMI≤24 (BMI= weight (kg)/height 2 (m2));
4. Complete physical examination: vital signs, hematuria routine, blood pregnancy, blood glucose, blood lipid,Blood electrolyte, hepatitis b surface antigen, liver and kidney function, hepatitis c, HIV and syphilis antibody test, Electrocardiogram, smoke test, urine drug screening, alcohol breath test, abdominal ultrasound examination, chest X-ray examination No abnormal or abnormal clinical significance;
5. Detailed understanding of the nature, significance, possible benefits and possible disadvantages of the experiment has been obtained before the study I was able to communicate well with the researchers, Comply with the requirements of the entire study and be able to understand and sign written informed consent.

Exclusion Criteria:

1. Have participated in any other clinical trials within the first three months of the trial;
2. Any diseases that may affect the safety of the test or the process of the drug in vivo, including But not limited to: heart, liver, kidney, endocrine, digestive tract, immune system and respiratory system Those with or existing diseases of the above system (especially those with cardiovascular diseases including cardiovascular diseases) Any gastrointestinal disease that affects drug absorption (such as irritable bowel syndrome symptoms, inflammation) History of sexual bowel), active pathological bleeding (such as peptic ulcer), urticaria, epilepsy, past Allergic rhinitis, eczema dermatitis, asthma, etc.
3. (consultation) allergy: if there are two or more drugs, food allergies or lactose intolerance Tolerance;
4. (consultation) any inhibition or induction of liver administration during the first 28 days of administration of the study drug Drugs for metabolism (common liver enzyme inducers: barbiturates Drugs for metabolism (common liver enzyme inducers: barbiturates such as phenobarbital, carbamazepine,Aminorumide, griseofulvin, aminopropyl, phenytoin, gluconate, rifampicin, desicer Betamethasone. Common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chlorine Mycin, isoniazid, sulfonamide, etc. Or had used any medication (pack) within 14 days prior to initial administration Including Chinese herbal medicine and health products;
5. (consultation) have specific food requirements and cannot follow a uniform diet (such as standard meals or high fat) Food intolerance) or difficulty swallowing;
6. (consultation) unable to tolerate venipuncture and/or having a history of blood or acupuncture;
7. (consultation) long-term overconsumption of tea and coffee (more than 8 cups a day, 1 cup =250mL) A person who drinks coffee or caffeine; Or 48 hours before the study's first dose Foods or drinks with caffeine (such as coffee, strong tea, chocolate, etc.) affect the absorption of drugs, A special diet of distribution, metabolism, and excretion;
8. (consultation) previous binge drinking (i.e., drinking more than 28 units per week for men and more than 28 units per week for women Drink more than 21 units of alcohol (1 unit contains 14 grams of alcohol, such as 360 mL of beer or 45 mL spirits of 40% alcohol or 150 mL wine); Or within 6 months prior to the trial Regular drinkers (more than 14 units per week); Or 24 before the first dose of the study Who has taken any alcoholic product within an hour;
9. (consultation) study blood donation or massive bleeding (greater than 450 mL) within 3 months before initial administration. Or who plans to donate blood or blood components during or within 3 months after the study;
10. (consultation) acute illness during the screening phase before study or before study medication;
11. (consultation) study of patients with liver replacement containing drugs that induce or inhibit liver replacement within 24 hours before initial administration Foods or drinks containing enzymes (e.g., grapefruit, mango, pitaya, grape juice, orange juice, etc.) are abundant Rich in flavonoids or citrus glycosides);
12. Surgery was performed within three months prior to the screening period or was planned for the duration of the study Surgery;
13. (consultation) previous history of drug abuse; A history of drug abuse;
14. (consultation) smoking more than 5 cigarettes per day during the 14 days before screening, or during the trial Using any tobacco products;
15. Screening of persons who have smoked or used any tobacco products up to admission;
16. Positive results of nicotine test;
17. Alcohol breath test with test results greater than 0.0mg/100ml;
18. Positive urine drug screening;
19. Pregnant women or those who plan to become pregnant within 6 months after the end of the trial;
20. The investigator considers that there is anything that may affect the subject's informed consent or adherence to the protocol Or participating in the test may affect the results of the test or the safety of the personnel under test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentration | up to 12 weeks
  Plasma drug concentration after administration of different doses of hydronidone

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics committee of drug clinical trials of huazhong university of science and technology, Wuhan, Hubei, China